CLINICAL TRIAL: NCT00753753
Title: Evaluation of the Occurence of Thrombotic and Bleeding Events After Coronary Angioplasty With Stent According to Aspirin and Clopidogrel Platelet Reactivity Assessed by a Point of Care Assay in the Cathlab (the Verifynow French Registry)
Brief Title: VerifyNow French Registry
Acronym: VERIFRENCHY
Status: Completed | Type: Observational
Sponsor: Association Pour le Développement des Soins Cardiologiques de la ville de Chartres (Other)
Collaborators: Medtronic (Industry); Boston Scientific Corporation (Industry); Cordis US Corp. (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, RANGE Gregoire, MD, Association Pour le Développement des Soins Cardiologiques de la ville de Chartres
Other Study IDs: VERIfynow FRENCH registrY; CPP n°2008-N2; AFFSAPS 2008-A00411-54
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Stent Thrombosis; Clopidogrel; Aspirin; Bleeding; Angioplasty
Keywords: stent thrombosis; clopidogrel; aspirin; bleeding; coronary; angioplasty
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the effect of clopidogrel or aspirin reactivity as measured by a point-of-care platelet function assay on thrombotic or bleeding events after percutaneous coronary intervention (PCI) with drug eluting or bare metal stent.

Methods:

Platelet reactivity on clopidogrel and aspirin therapy is measured before PCI with VerifyNow (Accumetrics Inc.,San Diego, CA, USA) P2Y12 or aspirin assay respectively in 1000 consecutive patients from 20 centers in France undergoing coronary angioplasty with stent.

Exclusion criteria are:

Acute myocardial infarction, treatment with vitamin K antagonists and the use of antiGP2b3a before PCI. All patients are pre-treated with clopidogrel and aspirin. Non-response to aspirin or clopidogrel is determined according to the result of the VerifyNow assay (cut off : < 15 % for P2Y12 and > 550 ARU for aspirin). The primary end point is the occurrence of definite or probable stent thrombosis (ARC definition) and the secondary end-points include global and cardio-vascular mortality, non fatal myocardial infarction and major bleeding. A clinical evaluation is scheduled at discharge and by telephone contact at one month and one year.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angioplasty with stent

Exclusion Criteria:

* Use of AGP2b3a
* Acute myocardial infarction
* No aspirin and clopidogrel pretreatment
* Use of AVK
* Aspirin or clopidogrel contre-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: real world patient referred for coronary angioplasty with stent
Sampling Method: Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Stent thrombosis | one year

SECONDARY OUTCOMES:
Mortality, cardio-vascular mortality, non fatal Myocardial infarction, urgent coronary revascularisation , re-hospitalization, severe bleeding | one year

CONTACTS AND LOCATIONS:
Overall Officials: gregoire rangé, Principal Investigator — GACI
Locations (1):
- cardiology unit / Les hopitaux de Chartres, Chartres, Eure Et Loir, France

REFERENCES:
- [Derived] Range G, Yayehd K, Belle L, Thuaire C, Richard P, Cazaux P, Barbou F, Koning R, Chassaing S, Teiger E, Berthier R, Decomis MP, Claudel JP, Delarche N, Brunel P, De Poli F, Dupouy P, Beygui F, Albert F, Collet JP, Montalescot G; VERIFRENCHY investigators. Thrombotic and bleeding events after coronary stenting according to clopidogrel and aspirin platelet reactivity: VerifyNow French Registry (VERIFRENCHY). Arch Cardiovasc Dis. 2014 Apr;107(4):225-35. doi: 10.1016/j.acvd.2014.03.004. Epub 2014 Apr 29. PMID 24794216